Assessment of Safety of Air Travel in Patients With Pulmonary Langerhans Cell Histiocytosis

NCT03052101

Document date: Feb. 23, 2017

Research Protocol

## **PLCH Survey**

You have been invited to participate in this research project because you have been diagnosed with Pulmonary Langerhans Cell Histiocytosis (PLCH).

This research project is being conducted by investigators in the Rare Lung Disease Consortium, a NIH funded organization consisting of multiple physicians and scientists dedicated to improving outcomes in rare lung diseases. This project is led by Dr. Abhishek Singla. The purpose of this research project is to gather information on lung collapse (pneumothorax) and the safety of air travel in patients with PLCH. In addition we aim to establish a contact registry to try to answer subsequent questions through this network of patients.

The procedure involves filling out an online survey that will take approximately 15 minutes. Your responses will be confidential, and you may choose to skip any questions that you do not want to answer, including your name and contact information if you wish to remain anonymous. If you choose provide it, your name and contact information will not be included in our data analyses. Although your participation in this research may not benefit you personally, it will help us understand how people live with PLCH, and guide future research directions.

Your participation in this research study is voluntary and you can choose not to participate. You can withdraw at any time even if you decide to participate in this research project. If you decide that you do not want to complete this survey, just close your browser.

We will do all we can to maintain confidentiality of your data. In order to keep your information confidential, all data is stored in a password protected electronic format in REDCap--an online data management system designed to protect research data. The clinical information collected for this study will be stored in a computer database at the University of Cincinnati (UC), the Cincinnati Children's Hospital Medical Center (CCHMC) and a federal data repository at the University of South Florida in Tampa, FL. A data repository provides a way for researchers to store the information collected during the research study for future research studies. The data management center at CCHMC and UC use several layers of protection for the clinical data stored in its computer database. It meets all of the local and federal security requirements for research datacenters. Your information is stored only using a study ID.

If you have any questions or concerns about participating in this project, please contact Elizabeth Kopras at koprasej@uc.edu or 513-558-7205.

Please call the University of Cincinnati Medical Institutional Review Board at 513-558-5259 (Monday - Friday 8 am to 5 pm) if you:

 Have general questions about giving consent or your rights as a research participant in this research study.

| <ul> <li>Have questions, concerns, or complaints about the</li> <li>Cannot reach the research team or you want to taproject.</li> </ul> | |
|---|---|
| • Think the research has hurt you. | |
| To report complaints or concerns to an independent manner, please call the Research Compliance Hotlin | |
| Thank you, | |
| Abhishek Singla, MD | |
| ELECTRONIC CONSENT: Please select your choice below. | <ul><li>○ Agree</li><li>○ Disagree</li></ul> |
| I would like to participate in this research study. | ) Disagree |
| Clicking on the "agree" button indicates that: • You have read the information above • You voluntarily agree to participate | |
| We request your permission to retain your name and contact information in a Patient Registry so that we can contact you for other studies. Rare diseases are difficult to study. Creating a Patient Registry will improve our ability to conduct research projects that can improve our understanding and management of PLCH. You can fill out this online survey without agreeing to participate in the Patient Registry. | <ul> <li>Yes, I agree that you may include my information in the Patient Registry, and contact me in the future to participate in other research studies.</li> <li>No, I do not want my information included in the Patient Registry. I do not want to be contacted for additional studies.</li> </ul> |
| I would prefer to be contacted by: | ☐ E-mail<br>☐ Telephone<br>☐ Regular mail |
| First Name<br>(optional) | |
| Last Name<br>(optional) | |
| Email address<br>(optional) | |
| Phone number (optional) | |
| Gender | <ul><li>○ Female</li><li>○ Male</li></ul> |
| Ethnicity | <ul><li>○ Hispanic</li><li>○ Non-Hispanic</li><li>○ Unknown</li><li>○ Prefer not to answer</li></ul> |

| Race | <ul> <li>Black or African American</li> <li>White or Caucasian</li> <li>American Indian or Alaska Native</li> <li>Native Hawaiian or Other Pacific Islander</li> <li>Asian</li> <li>Other</li> <li>Prefer not to answer</li> </ul> |
|---|---|
| Which of the following best describes your highest achieved education level? | <ul> <li>○ Graduate degree (Masters, Doctorate, etc.)</li> <li>○ Bachelor's degree</li> <li>○ Associate degree</li> <li>○ Some College, no degree</li> <li>○ High school graduate, no college</li> <li>○ Less than a high school diploma</li> </ul> |
| Date of Birth<br>(Please enter the date in Month/Day/Year format) | |
| PLCH HISTORY | |
| What was the approximate date when the symptoms or signs that you now know to be due to PLCH begin? - Please enter the date in Month/Day/Year format. | (If you don't remember the date, an estimate is fine.) |
| What was the approximate date that you were diagnosed with PLCH? (This could be before or after the start of your symptoms) | (If you don't remember the date, an estimate is fine.) |
| - Please enter the date in Month/Day/Year format. | |
| What was the first sign or symptom of PLCH that led to your diagnosis? (Check all that apply) | <ul> <li>No symptoms, was diagnosed on Chest X-Ray or CT scan incidentally</li> <li>Shortness of breath</li> <li>Cough</li> <li>Coughing up blood (hemoptysis)</li> <li>Collapsed lung (pneumothorax)</li> <li>Chest pain</li> <li>Fever</li> <li>Excessive sweating</li> <li>Weight loss (&gt; 10 percent of usual weight)</li> <li>Increased thirst or urination (Diabetes Insipidus)</li> <li>Bone lesions or bone pain</li> <li>Skin rash or lesions</li> <li>Enlarged lymph nodes</li> <li>Fatigue</li> <li>Other</li> </ul> |
| If you selected 'other', please specify: | |
| How long after your symptom onset were you diagnosed with PLCH? | <ul> <li>Less than 6 months</li> <li>6 months - 1 year</li> <li>1-2 years</li> <li>2-3 years</li> <li>3 years or more</li> <li>I had no symptoms before I was diagnosed</li> </ul> |



| How was your diagnosis of PLCH made?<br>(Check all that apply) | <ul> <li>☐ Chest X-ray</li> <li>☐ CT scan</li> <li>☐ Bronchoscopy</li> <li>☐ Lung Biopsy by surgery</li> <li>☐ Biopsy of other tissue, Please specify below</li> <li>☐ Other</li> </ul> |
|---|---|
| If you selected other, please specify: | |
| What manifestations of PLCH have you had, either past or present? (Check all that apply) | Cystic or bullous lung lesions (blebs) Personal history of pneumothorax (collapsed lung) Coughing up blood (hemoptysis) Chest pain Weight loss (> 10 percent of usual weight) Increased thirst or urination (Diabetes Insipidus) Pulmonary hypertension Bone lesions or bone pain Enlarged lymph nodes Fever, sweats, and/or chills Fatigue Other |
| If you selected other, please specify | |
| Prior to the correct diagnosis of PLCH, were you incorrectly diagnosed with a different disorder? | |
| If Yes, which incorrect diagnosis were you given | ☐ Asthma ☐ COPD or Emphysema ☐ LAM (Lymphangioleiomyomatosis) ☐ Lung Cancer ☐ Other ☐ Unsure/ Don't know |
| If you selected other, please specify | |
| BREATHING PROBLEMS | |
| Do you use supplemental oxygen for your symptoms? | |
| If yes, to what extent do you use supplemental oxygen? | <ul><li>Continuously</li><li>With exercise only</li><li>With sleep only</li><li>With sleep and exercise only</li></ul> |
| What is the flow rate (liters/minute) of supplemental oxygen that you usually use with activity? | |
| What is the flow rate (liters/minute) of supplemental oxygen that you usually use at rest? | |
| What is the flow rate (liters/minute) of supplemental oxygen that you usually use during sleep? | |



| Do you get short of breath with activity? | |
|---|---|
| The following best describes my shortness of breath? | <ul> <li>Not troubled by shortness of breath except with strenuous exercise</li> <li>Short of breath when hurrying on level ground or walking up a slight hill</li> <li>I walk slower than most people on the level, stop after a mile or so, or stop after 15 minutes when walking at my own pace</li> <li>I stop for breath after walking about 100 yards or after a few minutes on level ground</li> <li>I am too breathless to leave the house, or breathless when dressing</li> </ul> |
| Do you routinely use respiratory inhalers or bronchodilators? | |
| Besides PLCH what other lung problems do you have? (Check all that apply) | ☐ Asthma ☐ Pneumonia ☐ Emphysema/COPD ☐ Lung Cancer ☐ Other lung disease ☐ None |
| If you answered yes to 'Other diseases', please specify | |
| What other symptoms do you have from your lung disease? (Check all that may apply) | <ul><li>☐ Cough</li><li>☐ Coughing up blood</li><li>☐ Chest pain</li><li>☐ Other</li></ul> |
| If you selected other, please describe: | |
| Have you ever had a lung function test (PFT)? - This tests determine how much air your lungs can hold and how quickly you can move air in and out of your lungs. | <ul><li>Yes</li><li>Never had lung function testing</li><li>Unsure/Don't remember</li></ul> |
| How often do you have assessment of your lung function? | <ul> <li>Every 3 - 6 months</li> <li>Every 6 -12 months</li> <li>Every 1-2 years</li> <li>Less frequently than every two years</li> <li>Don't have regular lung function testing</li> <li>Unsure/Don't know</li> <li>Other</li> </ul> |
| If you selected other, please specify | |
| When was your last lung function test (PFT)? | |
| - Please enter the date in Month/Day/Year format. | (If you don't remember the date, an estimate is fine.) |

**₹EDCap**®

| What was your lung function (FEV-1) on your most recent test? | <ul><li>○ More than 80%</li><li>○ 50-80%</li><li>○ Less than 50%</li></ul> |
|---|---|
| FEV-1 is the Forced expiratory volume at timed intervals of 1.0 second | O Don't remember |
| SMOKING HISTORY | |
| Are you currently a cigarette smoker? | <ul><li>Yes</li><li>No</li></ul> |
| If not, did you smoke cigarettes in the past? | <ul><li>Yes- Quit</li><li>No- Never Smoked</li></ul> |
| If you smoke or used to smoke cigarettes, please estimate the number of years that you smoked? | |
| If you smoke or used to smoke cigarettes, how many cigarettes did you smoke in an average day? (1 pack= 20 cigarettes) | |
| When did you quit smoking cigarettes? | |
| - Please enter the date in Month/Day/Year format. | (If you don't remember the date, an estimate is fine.) |
| If you have quit smoking cigarettes, was there a reason that contributed to stopping smoking? Check all that apply. | <ul> <li>□ Pneumothorax (collapsed lung)</li> <li>□ Coughing up blood (hemoptysis)</li> <li>□ Shortness of breath</li> <li>□ Cost</li> <li>□ Concern about promoting disease progression</li> <li>□ Other</li> </ul> |
| If you selected 'Other' for the reason you quit smoking, please specify: | |
| What happened to your symptoms after quitting smoking? | <ul><li> Improved</li><li> Worsened</li><li> No Change</li></ul> |
| Was there a change in your Chest X-Ray or CT scan after you quit smoking? | <ul><li>Yes, improvement</li><li>Yes, worsening</li><li>No, stayed the same</li><li>Don't know/Not sure</li></ul> |
| Was there a change in your lung function after you quit smoking? | <ul><li>Yes, improvement</li><li>Yes, worsening</li><li>No, stayed the same</li><li>Don't know/Not sure</li></ul> |
| Do you smoke marijuana? | <ul><li>Yes, currently I smoke marijuana</li><li>Used to smoke in past but quit</li><li>No</li><li>Prefer not to answer</li></ul> |

| If you smoke or used to smoke marijuana, how often do or did you smoke? | <ul><li>Every day</li><li>1-2 times a week</li><li>1-2 times a month</li><li>Other</li></ul> |
|---|---|
| If you selected Other, please specify | |
| TREATMENT HISTORY | |
| Have you received any medication(s) other than inhalers for PLCH? | Yes No |
| If yes, please tell the name of the medication (check all that apply) | <ul> <li>☐ Chronic steroids directed at PLCH and not COPD (prednisone or Medrol)</li> <li>☐ Cladarabine (2-CDA)</li> <li>☐ Vemurafenib</li> <li>☐ Dabrafenib</li> <li>☐ Vincristine</li> <li>☐ Clofarabine</li> <li>☐ Cytarabine</li> <li>☐ Other</li> <li>☐ Don't know/Unsure</li> </ul> |
| If you selected Other, please specify other medications | |
| If you received PLCH treatment, what happened to your symptoms after treatment? | <ul><li>○ Improved</li><li>○ Worsened</li><li>○ No Change</li></ul> |
| If you received PLCH treatment, what happened to your Chest X-Ray or CT scan after treatment? | <ul><li>○ Improved</li><li>○ Worsened</li><li>○ No Change</li><li>○ Don't know/Not sure</li></ul> |
| If you recieved PLCH treatment, what happened to your lung function tests after treatment? | <ul><li>○ Improved</li><li>○ Worsened</li><li>○ No Change</li><li>○ Don't know/Not sure</li></ul> |
| Have you had a lung or a heart lung-transplant evaluation? | ○ Yes<br>○ No |
| Please check your current status. | <ul> <li>Being evaluated but not currently listed</li> <li>Listed for a lung or a heart lung-transplant</li> <li>Denied lung or a heart lung-transplant</li> <li>Undergone lung or a heart lung-transplant</li> </ul> |
| If you were not considered for lung transplant, what were the reason(s)? (check all that apply) | ☐ Active smoking ☐ Underweight or overweight ☐ Age ☐ Other medical reasons ☐ Other |
| Please specify your other reasons: | |

| If you have undergone transplant, please list the type of tran | splant and year it was done. |
|---|---|
| Right lung: Approximate date (M-D-Y) | |
| Left lung: Approximate date (M-D-Y) | |
| Both lungs: Approximate date (M-D-Y) | |
| Heart and Lung: Approximate date (M-D-Y) | |
| Where was the transplant done (which hospital)? | |
| FAMILY HISTORY | |
| Do you have family member(s) who also have PLCH ? (PLCH is not known to run in families) | <ul><li>Yes</li><li>No</li><li>Don't Know</li></ul> |
| If Yes, please specify the affected family member or members: (Check all that apply) | <ul> <li>Mother</li> <li>Father</li> <li>Sibling (s)</li> <li>Grandparent (s)</li> <li>Children</li> <li>Others</li> </ul> |
| If you selected Others, please specify: | |
| PNEUMOTHORAX (COLLAPSED LUNG) QUESTIONS | |
| Have you ever had a collapsed lung (pneumothorax)? | ○ Yes<br>○ No |
| If yes, how many episodes of pneumothorax have you had? | <ul> <li>○ 1</li> <li>○ 2</li> <li>○ 3</li> <li>○ 4</li> <li>○ 5</li> <li>○ 6</li> <li>○ More than 6</li> </ul> |

| What symptoms of pneumothorax (Check all that apply). | k did you experience? | <ul> <li>☐ Chest pain</li> <li>☐ Chest Pressure</li> <li>☐ Coughing up blood (Hemoptysis)</li> <li>☐ Shortness of Breath</li> <li>☐ Shoulder pain/back pain</li> <li>☐ Nausea</li> <li>☐ Dizziness</li> <li>☐ Unusual fatigue</li> <li>☐ Drop in oxygen saturation</li> <li>☐ Blue hands or nails</li> <li>☐ Anxiety</li> <li>☐ Other</li> <li>☐ None</li> </ul> | |
|---|---|---|---|
| Please specify your other sympton | ms: | | |
| Were you diagnosed with PLCH be of collapsed lung (pneumothorax) | | ○ Yes<br>○ No | |
| How many episodes of pneumoth to the diagnosis of PLCH? | orax did you have prior | <ul> <li>○ 1</li> <li>○ 2</li> <li>○ 3</li> <li>○ 4</li> <li>○ 5</li> <li>○ 6</li> <li>○ More than 6</li> </ul> | |
| For each episode of collaps and timing) | ed lung (pneumothora | x), please indicate the f | following (location |
| 1st Pneumothorax | Right | Left<br>( | Bilateral |
| 2nd Pneumothorax | $\circ$ | $\bigcirc$ | 0 |
| 3rd Pneumothorax | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| 4th Pneumothorax | 0 | 0 | 0 |
| 5th Pneumothorax | 0 | 0 | $\circ$ |
| 6th Pneumothorax | | | |
| | O | O | O |
| Date of first pneumothorax | | | |
| Date of first pneumothorax - Please enter the date in Month/D | Day/Year format. | (If you don't remember t | he date, an estimate is |
| · | Day/Year format. | | he date, an estimate is |
| - Please enter the date in Month/[ | | | |
| - Please enter the date in Month/D Date of second pneumothorax | | fine.) (If you don't remember t | |

06/21/2022 2:49pm

| Date of fourth pneumothorax | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| - Please enter the date in Month/Day/Year format. | | | | (If you don'<br>fine.) | t rememb | er the dat | e, an estima | te is |
| Date of fifth pneumothorax | | | | | | | | |
| - Please enter the date in Month/ | Day/Year fo | ormat. | | (If you don'<br>fine.) | t rememb | er the dat | e, an estima | te is |
| Date of sixth pneumothorax | | | | | | | | |
| - Please enter the date in Month/ | Day/Year fo | ormat. | | (If you don' fine.) | t rememb | er the dat | e, an estima | te is |
| Were you an active smoke | r (cigaret | tes and/ | or mariju | ana) at th | e time c | of the pr | eumothor | ax? |
| | Yes - Ciga | rettes Ye | s - Marijuana | Yes - E<br>cigarette<br>mariju | es and | No | Un | sure |
| 1st Pneumothorax | $\circ$ | | $\bigcirc$ | $\circ$ | | $\bigcirc$ | | $\circ$ |
| 2nd Pneumothorax | $\bigcirc$ | | $\bigcirc$ | $\circ$ | | $\bigcirc$ | 1 | $\circ$ |
| 3rd Pneumothorax | $\circ$ | | $\bigcirc$ | $\circ$ | | $\bigcirc$ | 1 | $\circ$ |
| 4th Pneumothorax | $\circ$ | | $\bigcirc$ | $\bigcirc$ | | $\bigcirc$ | $\circ$ | |
| 5th Pneumothorax | $\bigcirc$ | | $\bigcirc$ | $\bigcirc$ | | $\bigcirc$ | $\circ$ | |
| 6th Pneumothorax | 0 | | $\circ$ | 0 | | 0 | 0 | |
| What were you doing at th | e time yo | u had th | e pneum | othorax? | | | | |
| | Resting | Sleeping | Light work<br>/ Walking | Heavy<br>work /<br>Exercising | Flying | Deep<br>water<br>diving | Undergoin<br>g medical<br>procedure | Others |
| 1st Pneumothorax | | | | | | | | |
| 2nd Pneumothorax | | | | | | | | |
| 3rd Pneumothorax | | | | | | | | |
| 4th Pneumothorax | | | | | | | | |
| 5th Pneumothorax | | | | | | | | |
| 6th Pneumothorax | | | | | | | | |
| Please specify the medical proce applicable: | dure or oth | ers if | | | | | _ | |
| Did you have any of the fo | _ | | | | | | horax? | |
| | Neck or Ch | nest trauma | Air t | ravel | Deep wa | ter diving | Nor | ne |
| 1st Pneumothorax | [ | | [ | | [ | | | |
| 2nd Pneumothorax | [ | | [ | | | | | |
| | | | | | | _ | | |

06/21/2022 2:49pm

| 3rd Pneumothorax | | | | | | |
|---|---|---|---|---|---|---|
| 4th Pneumothorax | | | | | | |
| 5th Pneumothorax | | | | | | |
| 6th Pneumothorax | | | | | | |
| How was pneumothorax dia | | d many | CT C | | Oth | |
| 1st Pneumothorax | Chest > | k-ray<br> | CT Sc | an | Oth | er<br>] |
| 2nd Pneumothorax | | | | | | |
| 3rd Pneumothorax | | | | | | |
| 4th Pneumothorax | | | | | | |
| 5th Pneumothorax | | | | | | |
| 6th Pneumothorax | | | | | | |
| If Other, Please specify: | | | | | | |
| How long were you hospital | | | | | | |
| 1st Pneumothorax | Not hospitalized | < 1 day | 3-7 da | ıys 1-2 | weeks | > 2 weeks |
| 2nd Pneumothorax | | $\bigcirc$ | $\bigcirc$ | | | $\bigcirc$ |
| 3rd Pneumothorax | | $\bigcirc$ | $\bigcirc$ | | | $\bigcirc$ |
| 4th Pneumothorax | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | | $\bigcirc$ | $\bigcirc$ |
| 5th Pneumothorax | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | | $\bigcirc$ | $\bigcirc$ |
| 6th Pneumothorax | 0 | 0 | 0 | | 0 | 0 |
| How was each episode of your pneumothorax treated? (Please check all that apply for each episode) | | | | | | |
| Pleurodesis is a procedure i | n which the | lung is fuse | ed to the ch | est wall. Th | is can be do | one by |
| surgery (Surgical Pleurodes | | _ | ls such as t | alc, bleomy | cin, tetracy | cline or |
| povidone-iodine (called Che | | odesis).<br>Needle | Chest tube | Chaminal | Cumminal | Don't Know or |
| | Observation | aspiration | Chest tube | Chemical<br>Pleurodesis | Surgical<br>Pleurodesis | Unsure |
| 1st Pneumothorax | | | | | | |
| 2nd Pneumothorax | | | | | | |
| 3rd Pneumothorax | | | | | | |
| 4th Pneumothorax | | | | | | |
| 5th Pneumothorax | | | | | | |
| 6th Pneumothorax | | | | | | |



| If you had chemical pleuro | desis, what | type of che | mical was us | ed for the p | rocedure? | |
|---|---|---|---|---|---|---|
| | Talc | Bleomycin | | Povidone-lodi<br>ne | Other | Don't know /<br>unsure |
| 1st Pneumothorax | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| 2nd Pneumothorax | $\circ$ | $\circ$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\circ$ |
| 3rd Pneumothorax | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\circ$ | $\bigcirc$ | $\bigcirc$ |
| 4th Pneumothorax | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\circ$ | $\bigcirc$ | $\bigcirc$ |
| 5th Pneumothorax | $\circ$ | $\circ$ | $\circ$ | $\bigcirc$ | $\circ$ | $\circ$ |
| 6th Pneumothorax | 0 | 0 | 0 | 0 | 0 | 0 |
| Please specify if any other chem | ical was used | | | | | |
| FLIGHT HISTORY | | | | | | |
| Have you ever flown by airplane | ? | | ○ Yes | | | |
| | | | ○ No | | | |
| Are you a member of one or mor<br>programs | re airline frequ | ent flyer | ○ Yes ○ No | | | |
| How often do you fly, on average? | | | Once ev | ery 12 months<br>ery 6 months<br>ery 2-3 months<br>ery month | | |
| If other, please specify | | | | | | |
| Approximately how many flights you were diagnosed with PLCH? | have you take | n since | | | | |
| How many of these flights were | inter-continent | al? | | | | |
| Do you avoid air travel due to yo | our lung diseas | e? | ○ Yes<br>○ No | | | |
| Why do you avoid flying? | | | ☐ My own | n's advice<br>assessment of i<br>unrelated to m<br>asons | | |
| If you selected other above, plea | ase specify | | | | | |
| How has your flight frequency ch<br>diagnosed with PLCH? | nanged after yo | ou were | <ul><li>Increase</li></ul> | ge<br>ed frequency<br>d frequency<br>ely Stopped | | |

| Have you ever used supplementa | | ○ Yes<br>○ No | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Have you ever experienced any of the following during air travel (Developed only after getting on the flight)? (check all that apply) | | | | Shortness of breath Nausea Dizziness Chest pain Chest pressure Unusual fatigue Drop in oxygen saturation, by oximetry Headache Blue hands or nails Coughing up blood (Hemoptysis) Anxiety None of above | | | | |
| FLIGHT-RELATED PNEUMOT | HORAX | | | | | | | |
| We want to know if traveling pneumothorax (collapsed leftying and pneumothorax, afflights. Did you ever have a collapsed lunduring a flight or within a month of the collapsed lunduring afflight or within a month of the collapsed lunduring afflight or within a month of the collapsed lunduring afflight or within a month of the collapsed lunduring affigure of the collapsed lunduring affigu | and also | e followin<br>ask abou<br>othorax) | g questi<br>t your tr | ons ask | about rela | ationshi <sub> </sub> | ps betwee | |
| When do you feel that the | each of t | hese pne | umothor | ax happ | ened in re | elation t | o flight? | |
| | During a<br>flight | Within 24<br>hours of<br>flight | 1-2 days<br>after<br>flight | 3-7 days<br>after<br>flight | 1-2 weeks<br>after<br>flight | | | Don't<br>know |
| 1st Pneumothorax | $\circ$ | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| 2nd Pneumothorax | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| 3rd Pneumothorax | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| 4th Pneumothorax | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| 5th Pneumothorax | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\bigcirc$ | $\circ$ | $\bigcirc$ |
| 6th Pneumothorax | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 | $\circ$ |
| Please answer the followin | g questi | ons for fir | st flight | related | pneumotl | horax (d | uring or w | /ithin 2 |

| If you had a collapsed lung during a flight, what were the symptoms that you might have experienced? (Check all that apply). | ☐ Chest pain ☐ Chest Pressure ☐ Coughing up blood (Hemoptysis) ☐ Shortness of Breath ☐ Shoulder pain/back pain ☐ Nausea ☐ Dizziness ☐ Unusual fatigue ☐ Drop in oxygen saturation ☐ Blue hands or nails ☐ Anxiety ☐ Other | |
|---|---|---|
| If other, please specify | | |
| What specific kind of plane did you board when you had the first flight related pneumothorax? | <ul><li>Propeller plane</li><li>Small or Regional Jet</li><li>Large or Full sized Jet</li><li>Don't remember</li></ul> | |
| Please specify the boarding city of the flight on which this pneumothorax happened | | |
| Please specify the destination city of the flight on which this pneumothorax happened | | |
| How long was the flight that was associated with your pneumothorax (estimated hours)? | | |
| Was this a non-stop flight? | | |
| If no, how many connections did you make on that day? | <ul><li>○ 1</li><li>○ 2</li><li>○ 3</li><li>○ More than 3</li></ul> | |
| On which segment do you think the pneumothorax happened? | <ul><li> 1st</li><li> 2nd</li><li> 3rd</li><li> Other</li></ul> | |
| If other, please specify | | |
| At what point in the flight do you feel that your pneumothorax occurred? | <ul> <li>Prior to take off</li> <li>Ascending</li> <li>Cruise Altitude</li> <li>Descending</li> <li>After landing</li> </ul> | |
| Did you have any symptoms 24-48 hours prior to getting on the plane that were different from or worse than your usual symptoms of PLCH? | | |
| If yes, please describe | | _ |



| Was the flight crew aware you were having difficulty? Yes | Was PLCH diagnosed prior to the flight related pneumothorax? | ○ Yes ○ No |
|---|---|---|
| Oxygen supplementation Emergency plane landing Other Fother, please specify | Was the flight crew aware you were having difficulty? | |
| Were you hospitalized as a consequence of the flight related pneumothorax? Solution Solution | How were you managed on the plane? | <ul><li>Oxygen supplementation</li><li>Emergency plane landing</li></ul> |
| related pneumothorax? No | If other, please specify | |
| 1-2 days 3-7 days 1-2 weeks More than 2 weeks Chemical pleurodesis Chemical pleurodesis Surgical pleurodesis Other More than 2 weeks More than 3 w | | |
| Needle aspiration Chest tube Chemical pleurodesis Surgical pleurodesis Other | If yes, how many days did you stay in the hospital? | <ul><li> 1-2 days</li><li> 3-7 days</li><li> 1-2 weeks</li></ul> |
| OTHER QUESTIONS How many days after a pneumothorax were you told it was safe to fly? No recommendations given One day 1 week 2 weeks 1 month >1 month Old to avoid flying in the future Didnot have a pneumothorax Will you take flights in future? Yes No Only if it's an emergency | | <ul> <li>□ Needle aspiration</li> <li>□ Chest tube</li> <li>□ Chemical pleurodesis</li> <li>□ Surgical pleurodesis</li> </ul> |
| How many days after a pneumothorax were you told it was safe to fly? One day 1 week 2 weeks 1 month Told to avoid flying in the future Didnot have a pneumothorax Will you take flights in future? Yes No Only if it's an emergency | Please specify other treatments | |
| was safe to fly? One day 1 week 2 weeks 1 month Told to avoid flying in the future Didnot have a pneumothorax Will you take flights in future? Yes No Only if it's an emergency | OTHER QUESTIONS | |
| ○ No ○ Only if it's an emergency Is there anything else that you would like to tell us | | <ul> <li>One day</li> <li>1 week</li> <li>2 weeks</li> <li>1 month</li> <li>&gt;1 month</li> <li>Told to avoid flying in the future</li> </ul> |
| | Will you take flights in future? | ○ No |

| Have you reviewed your answers? |
|---|
| Scrolling may change your answers accidentally, depending on which internet browser you use. Please take a moment to review your answers before hitting the submit button below. |
| Thank you. |